CLINICAL TRIAL: NCT00547521
Title: A Phase IIIb, Multi-center, Stratified, Open-Label Study to Evaluate the Immunogenicity, Steady State Trough Level, and Safety of Subcutaneous Abatacept (BMS-188667) in Subjects With Rheumatoid Arthritis Administered With or Without Background Methotrexate
Brief Title: Phase IIIB Subcutaneous Abatacept Monotherapy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM101-173
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort (Experimental): In the ST period, participants were administered a dose of 125 mg abatacept SC, once weekly, for 4 months. Participants were also administered a stable MTX dose of greater than or equal to 10 mg once weekly for at least 4 weeks prior to first injection of SC abatacept.
  Interventions: Drug: abatacept; Drug: Methotrexate (MTX)
- SC Abatacept Monotherapy Cohort (Experimental): In the ST period, participants were administered a dose of 125 mg abatacept SC, once weekly, for 4 months. Participants did not receive MTX at screening i.e., MTX naive, or discontinued MTX due to lack of efficacy or tolerability at least 4 weeks prior to first injection of SC abatacept.
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept — solution, subcutaneous injection, 125 mg/kg, weekly, 106 days in short term; long term is open
  Other Names: BMS-188667; Orencia®
Drug: Methotrexate (MTX) — Participants who were currently receiving methotrexate at a stable dose ≥ 10 mg for at least 4 weeks
  Arms: Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort

SUMMARY:
To evaluate safety and immunogenicity of abatacept when used with or without methotrexate in the absence of an IV loading dose of abatacept

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rheumatoid Arthritis
* Subjects Global Disease Assessment of greater than equal to 20 mm on a visual analog scale
* Discontinue all Biologics and Disease-modifying antirheumatic drugs (DMARDS) except for methotrexate

Exclusion Criteria:

* Received treatment with rituximab
* Subjects who have received treatment with immunoadsorbtion columns (such as Prosorba columns), mycophenolate mofetil (Cellcept®), cyclosporine A or other calcineurin inhibitors, or D-Penicillamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (15):
  - Rheumatology Associates Of North Alabama, Huntsville, Alabama
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Stanford University School Of Medicine, Palo Alto, California
  - Boulder Medical Center, Boulder, Colorado
  - The Arthritis Center, Palm Harbor, Florida
  - Medical Towers South, Louisville, Kentucky
  - Westroads Medical Group, Omaha, Nebraska
  - Regional Rheumatology Associates, Binghamton, New York
  - Physicians East, Pa, Greenville, North Carolina
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - East Penn Rheumatology Associates, Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, Pa, Charleston, South Carolina
  - Columbia Arthritis Center, Columbia, South Carolina
  - Rheumatic Disease Center, Glendale, Wisconsin
- Australia (3):
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Hobart, Tasmania
  - Local Institution, Malvern, Victoria
- Mexico (2):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, D.f., Mexico City
- South Africa (2):
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape

REFERENCES:
- [Derived] Nash P, Nayiager S, Genovese MC, Kivitz AJ, Oelke K, Ludivico C, Palmer W, Rodriguez C, Delaet I, Elegbe A, Corbo M. Immunogenicity, safety, and efficacy of abatacept administered subcutaneously with or without background methotrexate in patients with rheumatoid arthritis: results from a phase III, international, multicenter, parallel-arm, open-label study. Arthritis Care Res (Hoboken). 2013 May;65(5):718-28. doi: 10.1002/acr.21876. PMID 23097311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Short term (ST) Study results (2 arms) were released in 2010. Final long term extension (LTE) results (1 arm with pooled data), up to 2014, are now included. During the LTE Study, 125 mg abatacept, was continued to be self-administered weekly and adjustments to RA medications including MTX were permitted at investigators discretion.
Pre-assignment Details: 119 participants enrolled;100 treated in the ST Study. Reasons not treated: 17 no longer met criteria, 2 withdrew consent. 96 completed ST treatment but only 95 completed Primary endpoint evaluation. 90 enrolled in LTE Study. Reasons why participants did not enroll in LTE Study: 2 lack of efficacy, 2 had adverse events, 1 no longer met criteria.
Groups:
- SC Abatacept Cohort: In the ST period, participants in this cohort were administered monotherapy, a dose of 125 mg abatacept SC, once weekly, for 4 months. Participants did not receive MTX at screening ie, MTX naive, or discontinued MTX due to lack of efficacy or tolerability at least 4 weeks prior to first injection of SC abatacept. During the LTE, all eligible participants continued to self-administer abatacept (125 mg SC) on a weekly basis with or without background MTX. During the LTE period, adjustments to RA medications (other than prohibited therapies), including MTX, were permitted at the investigator's discretion based upon the participant's clinical status. Consideration was given to decreasing corticosteroids and MTX in the presence of improvement in the participant's clinical condition. LTE period pooled all participants into 1 arm. Participation in the LTE continued until the abatacept SC formulation was commercially available in the country or until the study was terminated by the sponsor.
Period: Short Term Study (4 Months)
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Cohort
Started | 51 (Number of participants treated.) | 49 (Number of participants treated.)
Completed | 50 | 45
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal of consent | 0 | 1
Not completed — primary endpoint evaluation not complete | 0 | 1
Period: Long Term Extension (LTE) Study
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Cohort
Started | 0 (ST Study had 2 arms, LTE Study pooled all participants who had abatacept injection.) | 90 (ST Study had 2 arms, LTE Study pooled all participants who had abatacept injection.)
Completed | 0 | 59
Not Completed | 0 | 31
Not completed — Lack of Efficacy | 0 | 14
Not completed — Adverse Event | 0 | 9
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 0 | 2
Not completed — Poor/Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Median (Full Range); unit: years] | 55.0 (11.5) [34.0 to 84.0] | 54.0 (10.2) [26.0 to 68.0] | 54.0 (10.9) [26.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 41 | 75
  Male | 17 | 8 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 34 | 76
  Black | 7 | 4 | 11
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 1 | 10 | 11
  Other races | 0 | 1 | 1
Weight continuous [Mean (Standard Deviation); unit: kilogram (Kg)] | 84.6 (18.8) | 81.6 (22.4) | 83.1 (20.6)
Weight customized [Number; unit: participants]
  < 60 Kg | 4 | 8 | 12
  60 - 100 Kg | 36 | 31 | 67
  > 100 Kg | 11 | 10 | 21
Disease activity score C-reactive protein (DAS 28-CRP) [Mean (Standard Deviation); unit: Units on a scale] — DAS28-CRP is a continuous variable which is a composite of 4 variables: the number of tender joint out of 28, the number of swollen joint out of 28, C-reactive protein (CRP) in milligrams/Liter (mg/L) and participant assessment of disease activity measured on a visual analogue scale (VAS) of 100 millimeters (mm). DAS 28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * VAS + 0.96.
  Units on a scale | 5.1 (1.2) | 5.8 (1.5) | 5.4 (1.4)
Tender joints [Mean (Standard Deviation); unit: tender joints] — Total number of joints analyzed=68.
  tender joints | 23.9 (18.0) | 24.3 (14.2) | 24.1 (16.2)
Swollen joints [Mean (Standard Deviation); unit: swollen joints] — Total number of joints analyzed=66.
  swollen joints | 16.2 (12.0) | 18.3 (12.2) | 17.2 (12.1)
Subject pain assessment per Visual Analogue Scale(VAS) [Mean (Standard Deviation); unit: millimeters (mm)] — Subject Pain Assessment measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower value signifies a better Subject Pain Assessment.
  millimeters (mm) | 63.3 (19.1) | 70.5 (19.6) | 66.8 (19.6)
Subject global assessment per VAS [Mean (Standard Deviation); unit: mm] — Subject Global Assessment is measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower score indicates a better Subject Assessment of Global Health.
  mm | 60.4 (18.9) | 69.9 (22.6) | 65.0 (21.2)
Physician global assessment per VAS [Mean (Standard Deviation); unit: mm] — Physician Global Assessment is measured by VAS (100 mm). A Visual Analogue Scale (VAS) is a measurement instrument for characteristics that range across a continuum of values. Range is 1-100; a lower score indicates a better Physician Assessment of Global Health.
  mm | 51.6 (16.4) | 63.9 (20.5) | 57.7 (19.5)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: Units on a scale] — HAQ-DI takes into account participant's use of aids or devices or assistance in scoring algorithm for a disability category. The questionnaire includes 20 questions assessing physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty and 3 = unable to do. Higher scores indicate greater dysfunction. The score is calculated by summing worst scores in each domain and dividing by the number of domains answered.
  Units on a scale | 1.3 (0.7) | 1.5 (0.7) | 1.4 (0.7)
Rheumatoid Factor (RF) Status [Number; unit: participants] — RF is an autoantibody that is usually present in the serum of people with rheumatoid arthritis. The cut-point value for seroconversion was 15 International Unit (IU)/mL (>= 15 IU/mL resulted in a positive result).
  participants
    Unknown | 1 | 2 | 3
    Positive | 35 | 32 | 67
    Negative | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-abatacept or Anti-CTLA4-T Responses (Enzyme-linked Immunosorbent Assay [ELISA] Method) at Day 113 of the ST Study
Description: ELISA is a validated, sensitive assay technique used to analyze presence of abatacept-specific antibodies in serum. For anti-abatacept antibody ELISA, a sample was considered seropositive if it had a titer of 400 or greater and if immunodepletion was observed. The responses that were negative in initial screen were reported as seronegative with a value of < 400. A sample was considered positive in CTLA4-T antibody ELISA if it had a titer of 25 or greater and if immunodepletion was observed. The responses that were negative in initial screen were reported as seronegative with a value of < 25.
Time Frame: Day 113
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 50 | 45
participants | 0 | 0

2. Secondary Outcome: Change From Baseline in DAS28-CRP Score at End of 4-month (Day 113) of the ST Study
Description: DAS28-CRP is a continuous variable which is a composite of 4 variables: the number of tender joint out of 28, the number of swollen joint out of 28, C-reactive protein (CRP) in milligrams/Liter (mg/L) and subject assessment of disease activity measure on a VAS of 100mm. DAS 28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * VAS + 0.96.
Time Frame: Baseline and Month 4 (Day113).
Population: All treated participants included those participants who received at least 1 dose of the study medication (abatacept) in the ST period with baseline and post-baseline values.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 48 | 45
Units on a scale | -1.67 [-2.06 to -1.28] | -1.94 [-2.46 to -1.42]

3. Primary Outcome: Number of Participants With Anti-abatacept or Anti-CTLA4-T Responses (ELISA Method) Over Time During the ST Study
Description: as for outcome 1
Time Frame: Day 15, 29, 43, 57, 85,113 and 28, 56, and 85 days post last dose.
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses. n = those participants who were evaluated for this measure at each timepoint, for each group respectively.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Day 15, (n= 51,47) | 0 | 0
  Day 29, (n= 50,48) | 2 | 0
  Day 43, (n= 50,48) | 2 | 0
  Day 57, (n= 50,47) | 1 | 1
  Day 85, (n= 50,47) | 0 | 0
  Day 113, (n= 50,45) | 0 | 0
  Overall on Treatment visits, (n=51,49) | 2 | 1
  28 Days last post dose, (n=2,3) | 0 | 0
  56 Days last post dose, (n=2,3) | 0 | 0
  85 Days last post dose, (n=4,4) | 0 | 1
  Overall post visits, (n=4,4) | 0 | 1
  Overall, (n=51,49) | 2 | 2

4. Primary Outcome: Number of Participants With Positive Anti-abatacept Responses to Abatacept (Meso-Scale Discovery [MSD] Electrochemiluminescence [ECL] Assay Method) Over Time During the ST Study
Description: The ECL (MSD) assay method is a validated, sensitive assay technique used to analyze presence of abatacept-specific antibodies in serum. It is more sensitive and has a higher drug tolerance than ELISA method. For the anti-abatacept antibody ECL (MSD) assay, a sample was considered seropositive if it had a titer of 10 or greater and if immunodepletion was observed with abatacept, or abatacept and CTLA4-T. Those responses that were not positive in the initial screen or were not confirmed to be positive based on immunodepletion were reported as seronegative and were assigned a value of < 10.
Time Frame: Day 15, 29, 43, 57, 85,113 and 28, 56 and 85 days post last dose.
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses. n=number of participants who were evaluated for this measure at each timepoint, for each group respectively.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Day 15, (n= 51,47) | 1 | 1
  Day 29, (n= 50,48) | 1 | 0
  Day 43, (n= 50,48) | 1 | 0
  Day 57, (n= 50,47) | 1 | 0
  Day 85, (n= 50,47) | 1 | 0
  Day 113, (n=50,45) | 1 | 0
  Overall on Treatment visits, (n=51,49) | 1 | 1
  28 Days last post dose, (n=2,3) | 0 | 0
  56 Days last post dose, (n=2,3) | 0 | 0
  85 Days last post dose, (n=4,4) | 0 | 1
  Overall post visits, (n=4,4) | 0 | 1
  Overall, (n=51,49) | 1 | 2

5. Primary Outcome: Immunogenicity in MTX Naive and MTX-previous Users in Cohort 1 at Day 113 of the ST Study (for ELISA Results)
Description: as for outcome 1
Time Frame: Day 113.
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses. There were no positive Immunoglobulin G (IMG) samples on Day 113, therefore this analysis was not necessary.
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Immunogenicity in MTX Naive and MTX-previous Users in Cohort 1 at Day 113 of the ST Study (for MSD Results)
Description: The ECL (MSD) assay method is a validated, sensitive assay technique used to analyze presence of abatacept-specific antibodies in serum. It is more sensitive and has a higher drug tolerance than the ELISA method. For anti-abatacept antibody ECL (MSD) assay, a sample was considered seropositive if it had a titer of 10 or greater and if immunodepletion was observed with abatacept, or abatacept and CTLA4-T. Those responses that were not positive in the initial screen or were not confirmed to be positive based on immunodepletion were reported as seronegative and were assigned a value of < 10.
Time Frame: Day 113.
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses. There were no positive IMG samples on Day 113, therefore this analysis was not necessary.
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Cross Tabulations of the Number of Participants With Positive and Negative Immunogenicity Status at Baseline and Each Visit During the ST Study (for ELISA Results)
Description: as for outcome 1
Time Frame: Baseline and on day 15, 29, 43, 57, 85 and 113
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses.The overall percentage of subjects who had at least one positive sample was very low, therefore this analysis was not necessary.
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Cross Tabulations of the Number of Participants With Positive and Negative Immunogenicity Status at Baseline and Each Visit During the ST Study (for MSD Results)
Description: The ECL (MSD) assay method is a validated, sensitive assay technique used to analyze presence of abatacept-specific antibodies in serum . It is more sensitive and has a higher drug tolerance than the ELISA method. For anti-abatacept antibody ECL(MSD) assay, a sample was considered seropositive if it had a titer of 10 or greater and if immunodepletion was observed with abatacept, or abatacept and CTLA4-T. Those responses that were not positive in the initial screen or were not confirmed to be positive based on immunodepletion were reported as seronegative and were assigned a value of < 10.
Time Frame: Baseline and day 15, 29, 43, 57, 85 and 113.
Population: Treated participants in the ST period who were evaluable for anti-abatacept or anti-CTLA4-T responses. The overall percentage of subjects who had at least one positive sample was very low, therefore this analysis was not necessary.
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Meaningful Improvement at End of 4-month (Day 113) of the ST Study
Description: A clinically meaningful improvement is defined as a greater than or equal to 1.2 reduction in DAS28-CRP score from baseline.
Time Frame: Day 113.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 48 | 45
participants | 30 | 30

10. Secondary Outcome: Change From Baseline in Physical Functioning (HAQ-DI) at End of the 4-month Treatment Period (Day 113) of the ST Study
Description: HAQ-DI takes into account participant's use of aids or devices or assistance in scoring algorithm for a disability category. The questionnaire includes 20 questions assessing physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty and 3 = unable to do. Higher scores indicate greater dysfunction. The score is calculated by summing worst scores in each domain and dividing by the number of domains answered.
Time Frame: Baseline and Month 4 (Day 113).
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 49 | 46
Units on a scale | -0.31 [-0.43 to -0.19] | -0.58 [-0.74 to -0.42]

11. Secondary Outcome: Change From Baseline in All HAQ-DI Components at End of the 4-month Treatment Period (Day 113) of the ST Study
Description: as for outcome 10
Time Frame: Baseline and Month 4 (Day113).
Population: All treated participants included those participants who received at least 1 dose of the study medication (abatacept) in the ST period. n is the number of participants with baseline and post-baseline values.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
Units on a scale
  Dressing and Grooming, (n= 50,46) | -0.44 [-0.63 to -0.25] | -0.57 [-0.79 to -0.34]
  Arising, (n= 50,46) | -0.26 [-0.44 to -0.08] | -0.59 [-0.81 to -0.36]
  Eating, (n= 50,46) | -0.28 [-0.50 to -0.06] | -0.57 [-0.85 to -0.28]
  Walking, (n= 50,46) | -0.26 [-0.46 to -0.06] | -0.54 [-0.75 to -0.34]
  Hygiene, (n= 49,46) | -0.33 [-0.55 to -0.10] | -0.43 [-0.65 to -0.22]
  Reaching, (n= 49,46) | -0.24 [-0.47 to -0.02] | -0.50 [-0.74 to -0.26]
  Gripping, (n= 49,46) | -0.31 [-0.54 to -0.07] | -0.76 [-1.04 to -0.48]
  Activities, (n= 49,46) | -0.39 [-0.58 to -0.19] | -0.67 [-0.90 to -0.45]

12. Secondary Outcome: Cross Tabulations of Number of Participants With Positive and Negative Status for RF at Day 113 With Baseline, in the ST Study
Description: RF is an autoantibody that is usually present in the serum of people with rheumatoid arthritis. The cut-point value for seroconversion was 15 IU/mL (>= 15 IU/mL resulted in a positive result). Cross-tabulation of frequency of seroconversion of RF at Day 113 with baseline, in the ST period, was provided.
Time Frame: Baseline and Day 113.
Population: All treated participants included those participants who received at least 1 dose of the study medication (abatacept) in the ST period.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 47 | 45
participants
  Negative at Baseline, negative at Day 113 | 12 | 15
  Negative at Baseline, positive at Day 113 | 2 | 0
  Positive at Baseline, negative at Day 113 | 1 | 1
  Positive at Baseline, positive at Day 113 | 32 | 29

13. Secondary Outcome: Number of Participants Who Died, Experienced SAEs, Experienced AEs or Who Discontinued Due to AEs During the ST Study
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs or SAEs were recorded.
Time Frame: Continuously through ST period (upto Day 113). Includes the data from start of study drug therapy up to 56 days after the last dose (Day 113) or start of the long-term period whichever occurred first.
Population: All treated participants analysis population included all participants who received at least 1 dose of study medication (abatacept) in the ST period, were included in the safety analyses.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Deaths | 0 | 0
  SAEs | 2 | 3
  AEs | 37 | 32
  All SAEs Leading to Discontinuation | 1 | 1
  All AEs Leading to Discontinuation | 3 | 1

14. Secondary Outcome: Number of Participants Who Experienced Drug-related SAEs and Drug-related AEs During the ST Study
Description: Drug-related AEs are those events with a relationship to the study therapy of certain; probable; possible; or missing. Drug-related SAEs are those events with any relationship to the study therapy.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Drug-related AEs | 14 | 12
  Drug-related SAEs | 1 | 1

15. Secondary Outcome: Number of Participants With AEs of Special Interest During the ST Study
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). For this study, AEs of particular importance were associated with the use of immunomodulatory agents: infections, autoimmune disorders, malignancies, and injection reaction AEs (systemic AEs occurring within 24 hours of SC injection and local injection site reactions) were recorded.
Time Frame: Continuously through ST period (up to Day 113). Includes the data from start of study drug therapy up to 56 days after the last dose (Day 113) or start of the long-term period whichever occurred first.
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Infections | 18 | 14
  Malignant neoplasm | 0 | 0
  Autoimmune disorders | 0 | 0
  Local injection reactions | 3 | 4
  Systemic injection reactions | 4 | 4

16. Secondary Outcome: Number of Participants With Marked Abnormalities (MAs) in Hematology During the ST Study: Hemoglobin, Hematocrit, Platelet Count, Erythrocytes and Leukocytes
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Hemoglobin: >3 g/dL decrease from pre-treatment (pre Rx); hematocrit: <0.75 * pre-Rx value; platelet count: <0.67 * (LLN -lower limit of normal) (or, if pre-Rx value <LLN, then <0.5 * pre-Rx value and <100,000/mm^3); leukocytes: <0.75 * LLN or >1.25 * ULN (or, if pre-Rx value <LLN, then <0.8 * pre-Rx or >(ULN -upper limit of normal) ; erythrocytes: <0.75 * pre Rx.
Time Frame: Continuously from start of ST period up to 56 days post the last dose in the short-term period or start of the long-term period, whichever occurred first.
Population: All treated participants analysis population included all participants who received at least 1 dose of study medication (abatacept) in the ST period.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Low Hemoglobin | 0 | 0
  Low Hematocrit | 0 | 0
  Low Platelet Count | 0 | 0
  High Platelet Count | 0 | 0
  High Leukocytes | 1 | 2
  Low Erythrocytes | 0 | 0

17. Secondary Outcome: Number of Participants With MAs in Hematology During the ST Study: Neutrophils + Bands (Absolute), Lymphocytes (Absolute), Monocytes (Absolute), Basophils (Absolute) and Eosinophils (Absolute)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Neutrophils + bands (absolute): <1.00 * 10^3cells/microlitre (uL); lymphocytes (absolute): <0.75 * 10^3 cells/uL or >7.50 * 10^3 cells/uL; monocytes (absolute): >2.00 * 10^3 cells/uL; basophils (absolute): >0.40 * 10^3 cells/uL; eosinophils (absolute): >0.75 * 10^3 cells/uL.
Time Frame: as for outcome 16
Population: All treated participants analysis population included all participants who received at least 1 dose of study medication (abatacept)in the ST period.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  Low Neutrophils + Bands (absolute) | 0 | 0
  Low Lymphocytes (absolute) | 3 | 3
  High Lymphocytes (absolute) | 0 | 0
  High Monocytes (absolute) | 0 | 0
  High Basophils (absolute) | 0 | 0
  High Eosinophils (absolute) | 2 | 2

18. Secondary Outcome: Number of Participants With MAs in Serum Chemistry During the ST Study: Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Bilirubin (Total), G-Glutamyl Transferase (G-GT) and Blood Urea Nitrogen (BUN)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. ALP: >2.0 * ULN (if pre-Rx > ULN, then >3 * pre-Rx); AST, ALT: > 3 * ULN (if pre-Rx > ULN, then > 4 * pre-Rx); bilirubin (total): >2 * ULN, or if pre Rx > ULN then >4 * Pre Rx; BUN : >2 * pre Rx; GGT : >2 * ULN, or if pre Rx > ULN then >3 * pre Rx.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Number; unit: participants
Groups:
- Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort: In the ST period, participants were administered a stable MTX dose of greater than or equal to 10 mg once weekly for at least 4 weeks prior to first injection of SC abatacept. During LTE period, adjustments to MTX were permitted at the investigator's discretion based upon the participant's clinical status.
- SC Abatacept Monotherapy Cohort: In the ST period, participants were administered a dose of 125 mg abatacept SC, once weekly. Participants did not receive MTX at screening ie, MTX naive, or discontinued MTX due to lack of efficacy or tolerability at least 4 weeks prior to first injection of SC abatacept. During LTE period, all eligible participants continued to self administer abatacept (125 mg SC) on a weekly basis.
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  High ALP | 0 | 0
  High AST | 1 | 0
  High ALT | 1 | 0
  High GGT | 0 | 2
  High Bilirubin (total) | 0 | 0
  High BUN | 1 | 1

19. Secondary Outcome: Number of Participants With MAs in Serum Chemistry During the ST Study: Creatinine, Sodium (Serum), Potassium (Serum), Chloride (Serum), Calcium (Total) and Protein (Total)
Description: MAs= laboratory measurements marked as abnormal: creatinine: >1.5 * pre-Rx; sodium (serum):<0.95 * LLN or >1.05 * ULN (if pre-Rx < LLN, then <0.95 * pre-Rx or >1.05 * ULN. If pre-Rx > ULN, then >0.95 * pre-Rx or < ULN); potassium (serum):<0.9 * LLN or >1.1 * ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN; chloride (serum),protein (total):<0.9 * LLN or >1.1 8 ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN. If pre-Rx > ULN, then >1.1 * pre-Rx or < LLN); calcium (total): <0.8 * LLN or >1.2 * ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN. If pre-Rx > ULN, then >0.75 * pre-Rx or < ULN).
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  High Chloride (serum) | 0 | 0
  Low Chloride (serum) | 0 | 0
  High Calcium (total) | 0 | 0
  Low Calcium (total) | 0 | 0
  High Protein (total) | 0 | 0
  Low Protein (total) | 0 | 0
  High Creatinine | 0 | 1
  High Sodium (serum) | 0 | 0
  Low Sodium (serum) | 0 | 0
  Low Potassium (serum) | 1 | 0
  High Potassium (serum) | 0 | 0

20. Secondary Outcome: Number of Participants With MAs in Serum Chemistry During the ST Study: Glucose (Fasting Serum), Albumin, Glucose (Serum), Phosphorous (Inorganic) and Uric Acid
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following serum chemistry MA definitions specify MA criteria. Glucose (fasting serum): <0.8 * LLN or >1.5 ULN (if pre-Rx <LLN, then <2.0 * pre-Rx or >ULN; albumin: <0.9 * LLN (if pre-Rx < LLN, then <0.75 * pre-Rx); uric acid: >1.5 * ULN (if pre-Rx > ULN, then >2.0 * pre-Rx); phosphorous (inorganic):<0.75 * LLN or >1.25 * ULN (if pre-Rx < ULN, then <0.67 * pre-Rx or < ULN. If pre-Rx > ULN, then >1.33 * re-Rx or < LLN); glucose (serum): <65 mg/dL or >220 mg/dL.
Time Frame: as for outcome 16
Population: All treated participants analysis population included all participants who received at least 1 dose of study medication (abatacept) in the ST period, n= number of participants evaluated for this measure.
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  High Glucose (Fasting Serum) (n=8; n=21) | 0 | 0
  Low Glucose (Fasting Serum) (n=8; n=21) | 0 | 0
  Low Albumin (n=51; n=49) | 0 | 1
  Low Glucose (Serum) (n=51; n=49) | 6 | 1
  High Glucose(Serum) (n=51; n=49) | 2 | 1
  High Uric Acid (n=51; n=49) | 0 | 0
  High Phosphorous (inorganic) (n=51; n=49) | 0 | 0
  Low Phosphorous (inorganic) (n=51; n=49) | 1 | 1

21. Secondary Outcome: Number of Participants With MAs in Urinalysis During the ST Study: Protein, Glucose, Blood, Leukocyte Esterase, Red Blood Cells (RBC) and White Blood Cells (WBC)
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following definitions specify the criteria for MAs in urinalysis: protein, glucose, blood, leukocyte esterase, RBC, WBC: >= 2+ (or, if value >= 4, or if pre-Rx value = 0 or 0.5, then >= 2x or if pre-Rx value =1, then >= 3, or if pre-Rx = 2 or 3, then >= 4).
Time Frame: as for outcome 16
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants
  High Protein, urine (n= 51,49) | 0 | 2
  High Glucose, urine (n= 51,49) | 1 | 0
  High Blood, urine (n= 51,49) | 1 | 3
  High Leukocyte Esterase, urine (n= 18,17) | 2 | 3
  High WBC, urine (n= 15,19) | 3 | 6
  High RBC, urine (n= 12,17) | 1 | 7

22. Secondary Outcome: Number of Participants With Anti-nuclear Antibody (ANA) Category at Day 113 of the ST Study
Description: ANA status was categorized as negative or positive corresponding to the following dilutions: less than 1:160 and greater than equal to 1:160.
Time Frame: Day 113.
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 47 | 44
participants
  Negative | 36 | 32
  Positive | 11 | 12

23. Secondary Outcome: Number of Participants With Anti-double Stranded DNA (dsDNA) Category at Day 113 of the ST Study
Description: Anti-dsDNA antibody status was categorized as negative or positive based upon assay-specific numeric cut-off values.
Time Frame: Day 113.
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 45 | 45
participants
  Negative | 41 | 37
  Positive | 4 | 8

24. Secondary Outcome: Number of Participants With Clinically Meaningful Vital Signs During the ST Study
Description: Vital signs measurements (including seated blood pressure, heart rate and temperature) were recorded. The investigator used his/her clinical judgment to decide whether or not abnormalities in vital signs/physical examination were clinically meaningful.
Time Frame: At screening and on days 1,15,29,43, 57, 85 and 113.
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
participants | 0 | 0

25. Secondary Outcome: Minimum Plasma Concentration (Cmin) at Each Visit During the 4 Month Treatment Period of the ST Study
Description: Cmin serum abatacept concentration was obtained directly from the concentration-time data.
Time Frame: Days 1, 15, 29, 43, 57, 85 and 113.
Population: All treated participants analysis population included all participants who received at least 1 dose of study medication (abatacept) in the ST period. n=those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Geometric Mean (Full Range); unit: microgram/mL
Arm/Group | Subcutaneous (SC) Abatacept + Methotrexate (MTX) Cohort | SC Abatacept Monotherapy Cohort
Number analyzed (Participants) | 51 | 49
microgram/mL
  Day 15, (n= 40,41) | 13.69 [4.80 to 27.40] | 11.23 [2.70 to 27.10]
  Day 29, (n= 49,45) | 19.39 [6.10 to 41.80] | 15.64 [4.40 to 42.20]
  Day 43, (n= 41,38) | 23.40 [10.80 to 44.40] | 18.06 [5.20 to 48.10]
  Day 57, (n= 48,38) | 24.38 [10.90 to 41.10] | 21.71 [9.60 to 68.00]
  Day 85, (n= 47,39) | 28.77 [11.30 to 69.20] | 20.38 [2.60 to 50.00]
  Day 113, (n=46,37) | 28.46 [10.10 to 66.50] | 23.74 [6.60 to 70.80]

26. Secondary Outcome: Number of Participants With Abatacept Induced Antibody Responses Over Time During the LTE Study (ECL Method) - All Treated Participants in LTE Study
Description: The Meso-Scale Discovery (MSD) electrochemiluminescence (ECL) assay method is a validated, sensitive assay technique used to analyze presence of abatacept-specific antibodies in serum. It is more sensitive and has a higher drug tolerance than ELISA method. For the anti-abatacept antibody ECL (MSD) assay, a sample was considered seropositive if it had a titer of 10 or greater and if immunodepletion was observed with abatacept, or abatacept and CTLA4-T. Those responses that were not positive in the initial screen or were not confirmed to be positive based on immunodepletion were reported as seronegative and were assigned a value of < 10. Antibody responses included CTLA4 and possibly immune globulin (IG), IG and/or junction region.
Time Frame: Days 197, 281, 365, 449, 533, 617, 729, 813, 897, 981, 1093, 1177, 1261, 1345, 1457, 1541, 1625, 1709, 1821, 1989, days post dose: 28, 56, 85, 168
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had values at each specified timepoint, were evaluated.
Measure: Number; unit: participants
Groups:
- Abatacept Long Term Extension (LTE) Study: During the LTE Study, all eligible participants continued to self-administer abatacept (125 mg SC) on a weekly basis with or without background MTX. During the LTE Study, adjustments to RA medications (other than prohibited therapies), including MTX, were permitted at the investigator's discretion based upon the participant's clinical status. Consideration was given to decreasing corticosteroids and MTX in the presence of improvement in the participant's clinical condition. Participation in the LTE continued until the abatacept SC formulation was commercially available in the country or until the study was terminated by the sponsor.
Arm/Group | Abatacept Long Term Extension (LTE) Study
Number analyzed (Participants) | 90
participants
  Days 197, 281, 365, 449 (n=86, 87, 85, 79) | 0
  Day 533 (n=76) | 1
  Days 617, 729, 813 (n=74, 70, 66) | 0
  Days 897, 981 (n=66, 58) | 0
  Day 1093 (n=65) | 2
  Day 1177 (n=8) | 0
  Day 1261 (n=57) | 1
  Day 1345 (n=24) | 0
  Day 1457 (n=59) | 3
  Day 1541 (n=24) | 1
  Day 1625 (n=18) | 2
  Days 1709, 1821 (n=2, 11) | 0
  Day 1989 (n=13) | 1
  Overall on Treatment (n=88) | 11
  28 days post last dose (n=18) | 0
  56 days post last dose (n=15) | 2
  85 days post last dose (n=16) | 2
  168 days post last dose (n=3) | 2
  Overall post last dose visits (n=23) | 4
  Overall (n=90) | 13

27. Secondary Outcome: Change From Baseline in DAS28-CRP Score in the LTE Study - All Treated Participants in LTE Study
Description: DAS28-CRP is a continuous variable which is a composite of 4 variables: the number of tender joints out of 28, the number of swollen joints out of 28, C-reactive protein (CRP) in milligrams/Liter (mg/L) and subject assessment of disease activity measure on a VAS of 100mm. DAS 28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * VAS + 0.96. Baseline was Day 1 of the ST Study; Day 113 was the end of the ST Study.
Time Frame: Baseline, Day 113, Day 1345
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had DAS28-CRP values at Baseline, Day 113 and Day 1345, were evaluated.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Abatacept Long Term Extension Study: During the LTE Study, all eligible participants continued to self-administer abatacept (125 mg SC) on a weekly basis with or without background MTX. During the LTE Study, adjustments to RA medications (other than prohibited therapies), including MTX, were permitted at the investigator's discretion based upon the participant's clinical status. Consideration was given to decreasing corticosteroids and MTX in the presence of improvement in the participant's clinical condition.
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 88
Units on a scale
  Day 113 (n=88) | -1.89 [-2.2 to -1.5]
  Day 1345 (n=61) | -2.39 [-2.8 to -1.9]

28. Secondary Outcome: Number of Participants With Clinically Meaningful Improvement From Baseline in the LTE Study - All Treated Participants in LTE Study
Description: A clinically meaningful improvement is defined as a greater than or equal to 1.2 reduction in DAS28-CRP score from baseline. Baseline was Day 1 of the ST Study. Day 113 was the end of the ST Study.
Time Frame: Baseline, Day 113, Day 1345
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had values at Baseline, Day 113 and Day 1345, were evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 88
participants
  Day 113 (n=88) | 59
  Day 1345 (n=61) | 43

29. Secondary Outcome: Number of Participants in DAS28-CRP Remission and Number of Participants With Low Disease Activity (LDA) in the LTE Study - All Treated Participants in the LTE
Description: DAS28-CRP remission was defined as DAS28-CRP less than 2.6 and LDA was defined as DAS28-CRP less than, equal to 3.2. End of ST Study was Day 113.
Time Frame: Day 113, Day 1345
Population: Participants who received at least 1 dose of abatacept in the LTE study and who had values at Day 113 and Day 1345, were evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  Remission at Day 113 (n=90) | 28
  Remission at Day 1345 (n=63) | 28
  LDA at Day 113 (n=90) | 45
  LDA at Day 1345 (n=63) | 37

30. Secondary Outcome: Change From Baseline in HAQ-DI in the LTE Study - All Treated Participants in LTE Study
Description: HAQ-DI takes into account participant's use of aids or devices or assistance in scoring algorithm for a disability category. The questionnaire includes 20 questions assessing physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The questions are evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty and 3 = unable to do. Higher scores indicate greater dysfunction. The score is calculated by summing worst scores in each domain and dividing by the number of domains answered. Baseline was Day 1 in the ST Study and Day 113 was the last day of the ST Study.
Time Frame: Baseline, Day 113, Day 1345
Population: as for outcome 28
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 89
units on a scale
  HAQ-DI at Day 113 (n=89) | -0.47 [-0.57 to -0.36]
  HAQ-DI at Day 1345 (n=64) | -0.56 [-0.71 to -0.42]

31. Secondary Outcome: Number of Participants With HAQ Responses in the LTE Study - All Treated Participants in the LTE STudy
Description: HAQ response was defined as an improvement of at least 0.3 units from baseline in the HAQ Disability Index (HAQ DI). Baseline was Day 1 of the ST Study and Day 113 was the last day of the ST Study.
Time Frame: Baseline, Day 113, Day 1345
Population: as for outcome 28
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 89
participants
  HAQ DI Response at Day 113 (n=89) | 53
  HAQ DI Response at Day 1345 (n=64) | 41

32. Secondary Outcome: Number of Participants With Negative Status for RF up to 7 Days After Last Dose of Abatacept in the LTE Period - All Treated Participants in LTE Study
Description: RF is an autoantibody that is usually present in the serum of people with rheumatoid arthritis. The cut-point value for seroconversion was 15 IU/mL (>= 15 IU/mL resulted in a positive result).
Time Frame: Continuously from start of LTE period up to 7 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE and who had an RF test result up to 7 days post the last dose of abatacept in the LTE study, were evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 79
participants | 20

33. Secondary Outcome: Change From Baseline in DAS28-CRP Score and Physical Function (HAQ-DI) Score in the LTE Study - Abatacept Monotherapy Subgroup
Description: Abatacept Monotherapy Subgroup consisted of participants who received SC abatacept and did not receive MTX in the ST and LTE Studies. DAS28-CRP: continuous variable which is a composite of 4 variables:number of tender joints out of 28, number of swollen joints out of 28, C-reactive protein (CRP) in mg/L and self assessment of disease activity measure on a VAS of 100mm. DAS 28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.36 * ln(CRP+1) + 0.014 * VAS + 0.96. HAQ-DI includes 20 questions assessing physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty and 3 = unable to do. Higher scores indicate greater dysfunction. The score sums worst scores in each domain and divides by the number of domains answered. Baseline was Day 1 of Short Term Study. Day 113 was the last day of the Short Term Study.
Time Frame: Baseline, Day 113, Day 1345
Population: Participants who received abatacept monotherapy (at least 1 dose of abatacept and no MTX) in the ST and LTE Studies and who had values at Baseline, Day 113, and Day 1345, were evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Abatacept Monotherapy Subgroup: Abatacept Monotherapy Subgroup was defined as those participants who received as at least 1 dose of abatacept and did not receive MTX in the ST and LTE Studies.
Arm/Group | Abatacept Monotherapy Subgroup
Number analyzed (Participants) | 32
units on a scale
  DAS-CRP at Day 113 (n=31) | -2.42 (0.29)
  DAS-CRP at Day 1345 (n=23) | -2.58 (0.30)
  HAQ-DI at Day 113 (n=32) | -0.60 (0.10)
  HAQ-DI at Day 1345 (n=25) | -0.65 (0.12)

34. Secondary Outcome: Number of Participants in DAS 28-CRP Remission and Low Disease Activity (LDA) in the LTE Study - Abatacept Monotherapy Subgroup
Description: Remission was defined as DAS 28-CRP < 2.6 and LDA was defined as DAS 28-CRP <= 3.2. End of ST Study was Day 113. Abatacept Monotherapy Subgroup was defined as those participants who received as at least 1 dose of abatacept and did not receive MTX in the ST and LTE Studies.
Time Frame: Day 113, Day 1345
Population: Participants who received abatacept monotherapy (at least 1 dose of abatacept and no MTX) in the ST and LTE Studies, and who had values at Day 113 and Day 1345, were evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Monotherapy Subgroup
Number analyzed (Participants) | 32
participants
  Remission at Day 113 (n=32) | 14
  Remission at Day 1345 (n=24) | 9
  LDA at Day 113 (n=32) | 18
  LDA at Day 1345 (n=24) | 13

35. Secondary Outcome: Number of Participants Who Died, Experienced Serious Adverse Events (SAEs), Adverse Events (AEs), or Discontinued Due to AEs and/or SAEs During the LTE Period - All Treated Participants in LTE Study
Description: AEs: any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Drug-related AEs/SAEs are those events with a relationship to the study therapy of certain; probable; possible; or missing.
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had events up to 56 days post the last dose of abatacept in the LTE period, were evaluated. Includes all deaths reported during the LTE including those that occurred greater than 56 days after the last dose.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  Deaths | 0
  SAEs | 34
  Related SAEs | 6
  Discontinued due to SAEs | 3
  AEs | 86
  Related AEs | 34
  Discontinued due to AEs | 8

36. Secondary Outcome: Number of Participants With AEs of Special Interest During the LTE Study - All Treated Participants in LTE Study
Description: as for outcome 15
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had events up to 56 days post the last dose of abatacept in the LTE Study, were evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  Infections | 69
  Autoimmune Disorders | 5
  Malignancies | 4
  Local Injection Site Reactions | 2
  Systemic Injection Reaction | 12

37. Secondary Outcome: Number of Participants With Marked Abnormalities (MAs) in Hematology During the LTE Period - All Treated Participants in LTE Study
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. The following hematology MA definitions specify the criteria for the data presented. Hemoglobin: >3 g/dL decrease from pre-treatment (pre Rx); hematocrit: <0.75 * pre-Rx value; platelet count: <0.67 * (LLN -lower limit of normal) (or, if pre-Rx value <LLN, then <0.5 * pre-Rx value and <100,000/mm^3); leukocytes: <0.75 * LLN or >1.25 * ULN (or, if pre-Rx value <LLN, then <0.8 * pre-Rx or >(ULN -upper limit of normal) ; erythrocytes: <0.75 * pre Rx. Neutrophils + bands (absolute): <1.00 * 10^3cells/microlitre (uL); lymphocytes (absolute): <0.75 * 10^3 cells/uL or >7.50 * 10^3 cells/uL; monocytes (absolute): >2.00 * 10^3 cells/uL; basophils (absolute): >0.40 * 10^3 cells/uL; eosinophils (absolute): >0.75 * 10^3 cells/uL.
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had specified laboratory values up to 56 days post the last dose of abatacept in the LTE Study, were evaluated. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  Low Hemoglobin (n=90) | 1
  Low Hematocrit (n=90) | 0
  Low Erythrocytes (n=90) | 0
  Low Platelet Count (n=89) | 0
  High Platelet Count (n=89) | 0
  Low Leukocytes (n=90) | 2
  High Leukocytes (n=90) | 5
  Low Neutrophils + bands | 0
  Low Lymphocytes (n=90) | 6
  High Lymphocytes (n=90) | 1
  High Monocytes (n=90) | 2
  High Basophils (n=90) | 0
  High Eosinophils (n=90) | 13

38. Secondary Outcome: Number of Participants With MAs in Serum Chemistry (Liver and Kidney Function) During the LTE Period - All Treated Participants in LTE Study
Description: MAs are laboratory measurements marked as abnormal, per pre-defined study criteria, at any study time point. Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Bilirubin (Total), G-Glutamyl Transferase (G-GT), Blood Urea Nitrogen (BUN) and Creatinine MA criteria: ALP: >2.0 * ULN (if pre-Rx > ULN, then >3 * pre-Rx); AST, ALT: > 3 * ULN (if pre-Rx > ULN, then > 4 * pre-Rx); bilirubin (total): >2 * ULN, or if pre Rx > ULN then >4 * Pre Rx; BUN : >2 * pre Rx; GGT : >2 * ULN, or if pre Rx > ULN then >3 * pre Rx; creatinine: >1.5 * pre-Rx.
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and with specified laboratory values up to 56 days post the last dose of abatacept in the LTE Study, were evaluated. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  High ALP (n=90) | 0
  High AST (n=90) | 1
  High ALT (n=90) | 3
  High G-GT (n=90) | 2
  High Bilirubin (n=90) | 0
  High BUN (n=90) | 6
  High Creatinine (n=90) | 7

39. Secondary Outcome: Number of Participants With MAs in Serum Chemistry (Electrolytes, Glucose, Protein, and Metabolite) During the LTE Period - All Treated Participants in LTE Study
Description: Sodium (serum):<0.95 * LLN or >1.05 * ULN (if pre-Rx < LLN, then <0.95 * pre-Rx or >1.05 * ULN. If pre-Rx > ULN, then >0.95 * pre-Rx or < ULN); potassium (serum):<0.9 * LLN or >1.1 * ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN; chloride (serum),protein (total):<0.9 * LLN or >1.1 8 ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN. If pre-Rx > ULN, then >1.1 * pre-Rx or < LLN); calcium (total): <0.8 * LLN or >1.2 * ULN (if pre-Rx < LLN, then <0.9 * pre-Rx or > ULN. If pre-Rx > ULN, then >0.75 * pre-Rx or < ULN); phosphorous (inorganic):<0.75 * LLN or >1.25 * ULN (if pre-Rx < ULN, then <0.67 * pre-Rx or < ULN. If pre-Rx > ULN, then >1.33 * re-Rx or <LLN); glucose (serum): <65 mg/dL or >220 mg/dL; Glucose (fasting serum): <0.8 * LLN or >1.5 ULN (if pre-Rx <LLN, then <2.0 * pre-Rx or >ULN; albumin: <0.9 * LLN (if pre-Rx < LLN, then <0.75 * pre-Rx); uric acid: >1.5 * ULN (if pre-Rx > ULN, then >2.0 * pre-Rx).
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had specified laboratory values up to 56 days post the last dose of abatacept in the LTE study, were summarized. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 90
participants
  High and/or Low Sodium (n=90) | 0
  Low Potassium (n=90) | 2
  High Potassium (n=90) | 0
  High and/or Low Chloride | 0
  High and/or Low Total Calcium (n=90) | 0
  High and/or Low Inorganic Phosphorus (n=90) | 0
  Low Glucose (n=90) | 21
  High Glucose (n=90) | 1
  Low Fasting Glucose (n=28) | 3
  High Fasting Glucose (n=28) | 1
  High and/or Low Total Protein (n=90) | 0
  Low Albumin (n=90) | 0
  High Uric Acid (n=90) | 1

40. Secondary Outcome: Number of Participants With MAs in Urinalysis During the LTE Period: Protein, Glucose, Blood, Leukocyte Esterase, Red Blood Cells (RBC) and White Blood Cells (WBC) - All Treated Participants in LTE Study
Description: as for outcome 21
Time Frame: Continuously from start of LTE Study up to 56 days post the last dose
Population: Participants who received at least 1 dose of abatacept in the LTE Study and who had specified laboratory values up to 56 days post the last dose of abatacept in the LTE period, were evaluated. n=number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Abatacept Long Term Extension Study
Number analyzed (Participants) | 89
participants
  High Urine Protein (n=89) | 6
  High Urine Glucose (n=89) | 2
  High Urine Blood (n=89) | 13
  High Urine Esterase (n=45) | 12
  High Urine WBC (n=51) | 26
  High Urine RBC (n=47) | 16

ADVERSE EVENTS:
Time Frame: Short Term (ST) Study: Day 1 up to Day 113. LTE Study: Start of LTE Study up to 56 days post the last dose. Study initiated 2007 and completed LTE 2014.
Description: ST: includes data from start of study drug therapy up to 56 days after the last dose (Day 113) or start of the long-term period whichever occurred first. Participants could enter LTE at the conclusion of the ST and could continue in the LTE until the SC formulation was commercially available or until the study was terminated by the sponsor.
Groups:
- Short Term Study: Subcutaneous (SC) Abatacept + Methotrexate: In the ST period, participants were administered a dose of 125 mg abatacept SC, once weekly, for 4 months. Participants were also administered a stable MTX dose of greater than or equal to 10 mg once weekly for at least 4 weeks prior to first injection of SC abatacept.
- Short Term Study: SC Abatacept Monotherapy: In the ST period, participants were administered a dose of 125 mg abatacept SC, once weekly, for 4 months. Participants did not receive MTX at screening i.e., MTX naive, or discontinued MTX due to lack of efficacy or tolerability at least 4 weeks prior to first injection of SC abatacept.
- Long Term Extension (LTE):125 mg SC Abatacept: During the LTE Study, all eligible participants continued to self-administer abatacept (125 mg SC) on a weekly basis with or without background MTX. During the LTE Study, adjustments to RA medications (other than prohibited therapies), including MTX, were permitted at the investigator's discretion based upon the participant's clinical status. Consideration was given to decreasing corticosteroids and MTX in the presence of improvement in the participant's clinical condition.
Arm/Group | Short Term Study: Subcutaneous (SC) Abatacept + Methotrexate | Short Term Study: SC Abatacept Monotherapy | Long Term Extension (LTE):125 mg SC Abatacept
Serious Adverse Events (participants affected / at risk) | 2/51 | 3/49 | 34/90
Other Adverse Events (participants affected / at risk) | 16/51 | 13/49 | 70/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Short Term Study: Subcutaneous (SC) Abatacept + Methotrexate (N=51) | Short Term Study: SC Abatacept Monotherapy (N=49) | Long Term Extension (LTE):125 mg SC Abatacept (N=90)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 2
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gliosis (Nervous system disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 1 | 0 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Short Term Study: Subcutaneous (SC) Abatacept + Methotrexate (N=51) | Short Term Study: SC Abatacept Monotherapy (N=49) | Long Term Extension (LTE):125 mg SC Abatacept (N=90)
Pneumonia (Infections and infestations) | 0 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Fatigue (General disorders) | 0 | 0 | 5
Insomnia (Psychiatric disorders) | 0 | 0 | 6
Sinusitis (Infections and infestations) | 0 | 0 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Depression (Psychiatric disorders) | 0 | 0 | 5
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 8
Hypertension (Vascular disorders) | 0 | 0 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 0 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 2 | 21
Cellulitis (Infections and infestations) | 0 | 0 | 5
Bronchitis (Infections and infestations) | 0 | 0 | 12
Headache (Nervous system disorders) | 5 | 3 | 5
Influenza (Infections and infestations) | 0 | 0 | 7
Nasopharyngitis (Infections and infestations) | 0 | 0 | 12
Gastroenteritis (Infections and infestations) | 0 | 0 | 5
Tooth abscess (Infections and infestations) | 0 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 8
Herpes zoster (Infections and infestations) | 0 | 0 | 7
Urinary tract infection (Infections and infestations) | 1 | 3 | 17
Vomiting (Gastrointestinal disorders) | 0 | 4 | 0
Injection site pruritus (General disorders) | 3 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period <= 60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.